CLINICAL TRIAL: NCT05159427
Title: Open-Label, Randomized, Pharmacokinetic Study of Single-Dose Modified Release Glipizide in Healthy Volunteers
Brief Title: Pharmacokinetic Study of Single-Dose Modified Release Glipizide in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Duxin Sun, Charles R. Walgreen Jr. Professor of Pharmacy and Professor of Pharmaceutical Sciences, College of Pharmacy, The University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00199603
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Human Gastrointestinal Physiology Data
Keywords: Clinical study; Glipizide; Modified release; Pharmacokinetics; In vivo dissolution; Local gastrointestinal concentration
MeSH Terms: interventions — Glipizide; Rifaximin

STUDY DESIGN:
Intervention Model Description: This is a parallel study design. Subjects are asked to complete the study events/procedures in one phases (G.I intubation) with one of the two formulations of glipizide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- G.I Intubation (Experimental): Single dose of Glipizide (5 mg modified-release tablet) and Rifaximin (200 mg tablet) administered with 200 mL of 20% glucose solution in water + 1 mg of the stable isotope Glipizide (13C6-Glipizide) with 40 ml of 14% glucose solution in water. A 'Stable isotope' means a heavier version of the drug that is not radioactive.
  Interventions: Drug: Glucotrol XL 5Mg Extended-Release Tablet; Drug: Glipizide ER 5 MG 24 HR Extended Release Oral Tablet; Drug: Rifaximin 200Mg Tab; Drug: 13C6-Glipizide

INTERVENTIONS:
Drug: Glucotrol XL 5Mg Extended-Release Tablet — Participants are randomized to take one tablet of this study drug by mouth.
Drug: Glipizide ER 5 MG 24 HR Extended Release Oral Tablet — Participants are randomized to take one tablet of this study drug by mouth.
Drug: Rifaximin 200Mg Tab — Participants will take one tablet of this study drug by mouth.
Drug: 13C6-Glipizide — Participants will take 1 mg of this study drug dissolved in 40 ml glucose solution by mouth.
  Other Names: Stable Isotope Glipizide

SUMMARY:
In vivo drug dissolution in the gastrointestinal (GI) tract is largely unmeasured. The purpose of this clinical study is to evaluate the in vivo drug dissolution and systemic absorption of modified release formulations of the BCS Class II drug Glipizide by direct sampling of stomach and small intestinal luminal content, blood, urine and feces.

Expanding current knowledge of drug dissolution in vivo will help to establish physiologically relevant in vitro models predictive of drug dissolution.

DETAILED DESCRIPTION:
This is an in vivo study designed to acquire human gastrointestinal (GI) physiology data from healthy subjects which are necessary for mechanistic absorption model development. Each subject will be asked to complete a single dosing phase. The dosing phase will include collection of fluids from stomach and gastrointestinal (GI) tract through intubation (putting a GI tube from mouth into stomach and intestines), blood, urine and feces, and measure glipizide concentrations.

The objectives of this study are, as follows: Objective #1: To characterize the plasma, gastrointestinal fluid, urine, and feces concentrations of glipizide after oral administration of modified release formulations; Objective #2: To compare the pharmacokinetics of glipizide between the two modified release formulations; Objective #3: To collect gastrointestinal physiology data in volunteers receiving an oral MR formulation of glipizide. These in vivo results will be used to validate in vitro dissolution methods and to support computational and mathematical modeling efforts, in order to develop an oral drug product optimization process that may be applied to future drugs to maximize oral drug safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults age 18 to 55 years with BMI ranging from 18.5 to 35 kg/m2 inclusive
2. Ability to independently provide an informed consent
3. Demonstrate the ability to swallow a multivitamin pill that mimics a SmartPill capsule
4. Negative serum pregnancy test (for women of child-bearing potential)

Exclusion Criteria:

1. Unable to independently provide an informed consent for themselves or mentally incapacitated.
2. Physical disability (including blindness or deafness) that requires special arrangements.
3. Significant clinical illness, including cardiovascular disease, neurological disease, organ failure, or malignancy in the opinion of the investigator
4. Any surgical procedure within 3 weeks prior to screening
5. History and/or presence of severe seasonal allergies or severe allergic diseases including drug allergies, food allergies and allergy against the SmartPill® device
6. History and/or presence of hypersensitivity to any of the study drugs or the products' excipients
7. History and/or presence of hypersensitivity to Sulfonamide derivatives
8. History and/or presence of hypersensitivity to Lidocaine
9. History and/or presence of hypersensitivity to rifaximin, rifamycin antimicrobial agents, or any of the components of XIFAXAN
10. History and/or presence of hypersensitivity to acrylate or methacrylate, commonly used components of medical adhesives
11. Any other factor, condition, or disease, including, but not limited to, cardiovascular, respiratory, hematological, renal, hepatic, or gastrointestinal disorders that may, in the opinion of the Investigator, jeopardize the safety of the patient, alter drug absorption and pharmacokinetics or impact the validity of the study results.
12. Subjects with Type 1 Diabetes Mellitus (DM), diabetic ketoacidosis, with or without coma
13. Subjects with Glucose 6-phosphate dehydrogenase (G6PD) deficiency
14. History and/or presence of drug addiction or alcohol abuse within the past 12 months.
15. History of significant psychiatric or neurological illness, including seizure disorders.
16. Any medical or surgical conditions which might significantly interfere with the functions of gastrointestinal tract (e.g., gastric/intestinal bypass surgeries, fistulas, strictures, stenosis, or physiological/mechanical obstruction of the G.I tract, gastric bezoars, irritable bowel disease, crohn's disease, diverticulosis, or chronic narcotic use).
17. History of dysphagia to liquids, food, or pills
18. History of abdominal radiation therapy
19. Pregnant or lactating females
20. Any clinically significant abnormal lab values during screening in the opinion of the investigator.
21. Use of alcohol and/or nicotine containing products 48 hours prior to dosing visits, and throughout PK sampling visits.
22. Use of any medications and/or supplements, prescriptions or over the counter 1 week prior to beginning the study, and throughout the study except for birth control with approved methods of contraception when used consistently and correctly (Implants (i.e. Implanon, Nexplanon), Injectables (i.e. Depo-Provera), Combined, Oral Contraceptives, Intrauterine Devices (IUD's) (i.e. Mirena, ParaGard), and Sexual Abstinence are accepted).
23. Use of aspirin or any blood thinner medications.
24. Use of an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump.
25. Volunteers unwilling or unable to take the proposed drugs or undergo G.I intubation
26. Enrollment in a clinical trial in the past 30 days
27. Current enrollment in a clinical trial with another study drug, vaccine or medical device
28. Fasting blood glucose level < 80 mg/dL.
29. Inability or unwillingness to fast for 19 hours.
30. Blood donations in the past 8 weeks except for apheresis.
31. Volunteer shows a positive result of COVID-19 Antigen Rapid test in dosing visits
32. Volunteer is having any of the following symptoms:

    * Fever (over 100.4 oF or 38 oC) or feeling feverish
    * New cough
    * New shortness of breath
33. Volunteer is having two of any of these symptoms:

    * Chills
    * Muscle aches
    * New URI symptom(s) (runny nose, nasal congestion, and/or sore throat)
    * New loss of sense of smell or sense of taste
    * New headache
34. Volunteer has been in close contact in the last 14 days with someone recently diagnosed with COVID-19
35. Volunteer has returned from international travel within the past 10 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Average Area Under the Plasma Concentration-time Curve to infinite time (AUCinfinity) of Glipizide After a Single Dose of Glipizide with Gastrointestinal Intubation and between Two Modified Release Glipizide formulations | From time 0 to 78 hours
  Average Area Under the Plasma Concentration-time Curve to infinite time (AUCinfinity) of Glipizide will be measured at multiple timepoints over a 78 hour period at each of the two study phases

SECONDARY OUTCOMES:
Plasma Cmax of Glipizide After a Single Dose of Glipizide with Gastrointestinal Intubation and between Two Modified Release Glipizide formulations | From time 0 to 78 hours
  Peak Plasma Concentration of Glipizide (Cmax) will be measured at multiple timepoints over a 78 hour period at the study phase
Plasma Tmax of Glipizide After a Single Dose of Glipizide with Gastrointestinal Intubation and between Two Modified Release Glipizide formulations | From time 0 to 78 hours
  The time it takes to reach the maximum concentration of Glipizide in Plasma (Tmax) will be measured at multiple timepoints over a 78 hour period at the study phase
Urine and Feces concentrations of Glipizide After a Single Dose of Glipizide with Gastrointestinal Intubation and between Two Modified Release Glipizide formulations | From time 0 to 78 hours
  Recovery of Glipizide in urine and feces will be measured at multiple timepoints over a 78 hour period at the study phase
Maximum Gastrointestinal fluid concentration of Glipizide after Oral Administration of a Single Dose Modified Released Formulation of Glipizide | From time 0 to 7 hours
  The concentration of Glipizide in gastrointestinal fluid (stomach, duodenum, jejunum and ileum) will be measured at multiple timepoints over a 7 hour period using a 4-port G.I Intubation Catheter
Gastrointestinal pH after Oral Administration of Modified Release Formulation of Glipizide | From time 0 to 7 hours
  Gastrointestinal pH will be measured ex-vivo in gastrointestinal fluid samples collected through gastrointestinal intubation catheter over a duration of 7 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Ring, Study Director — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States